CLINICAL TRIAL: NCT04113044
Title: Clinical Priority Program (CPP) Clinical Outcome Measurement of Fracture Treatment:
Brief Title: Go Fit Fast, Recovery Trajectory Using PROMIS®, Linking PROMIS®
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: CPP Patient Outcome
Record Dates: First submitted 2019-09-20; First posted 2019-10-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hip Fractures; Tibial Fractures; Ankle Fractures; Humeral Fracture, Proximal; Distal Radius Fracture
Keywords: PRO; HOOS; KOOS; FAAM; PROMIS; QuickDASH; PSEQ; PAM
MeSH Terms: conditions — Hip Fractures; Tibial Fractures; Ankle Fractures; Shoulder Fractures; Wrist Fractures | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: All treatments will remain the standard (routine) care procedures based on individual clinician's judgment and the patient characteristics. — All treatments will remain the standard (routine) care procedures based on individual clinician's judgment and the patient characteristics.
  Other Names: Patient Reported Outcomes

SUMMARY:
Prospective data will be collected in approximately 3500 patients (700 per 5 injury groups).

Patients will be followed up according to the standard (routine) for up to 1 year after the treatment.

Data collection will include underlying disease, treatment details, patient reported outcomes (PROs), anticipated or procedure-related adverse events (i.e. complications), and radiological outcomes.

DETAILED DESCRIPTION:
More in detail this observational study includes the following sub-projects:

I) Weight -bearing and Gait Observation for Fully Individualized Treatment and Aftercare Following Surgery and Trauma

Objectives:

To analyse the association between automated, sensor-based patient activity and loading data, and clinical (Patient Reported Outcomes [PROs]) and radiographic outcome during fracture healing.

II) Recovery Trajectory using PROMIS®: Defining the Recovery Trajectory using PROMIS® to Optimize Decision-making and Outcomes following Extremity Fractures

Objectives:

1. To identify the factors predictive of longer term magnitude of limitations after extremity fractures (using PROMs)
2. To assess minimal clinically important difference (MCID) and substantial clinical benefit (SCB) in PROM scores
3. To define recovery trajectories of PROMs i.e. range, normative limits and score thresholds

III) Linking PROMIS®: Linking of PROMIS Measures to Legacy Measures in an Orthopaedic Patient Population

Objectives:

1. Administer and collect responses to the PROMIS PF/UE and PAIN INT and the four orthopaedic legacy measures in the same group of orthopaedic trauma patients.
2. Apply the methods of item-response theory (IRT) linking to establish a common standardized metric.
3. Develop equations for conversion of a PROMIS PF/UE and PAIN INT score to each of the specified legacy measures and vice-versa.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of one of, isolated injury

  * Hip fracture
  * Tibial shaft fracture (with and without associated fibular fracture)
  * Ankle/pilon fracture
  * Proximal humerus fracture
  * Distal radius fracture
* English, German, or Spanish speaking
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
  * Signed and dated EC/IRB approved written informed consent

Exclusion Criteria:

* More than 14 days from day of injury to day of surgery / day of nonoperative treatment decision
* Patients with multiple fractures
* Pathological fractures due to cancer
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the study period
* Patients who are not able to provide independent written informed consent unless defined and IRB/IEC-approved procedures for consenting such vulnerable patients are in place
* Prisoners
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study
* Patients unable to likely achieve anticipated Follow-up (FU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 who have have suffered an isolated fracture of one of the following five bones: 1. proximal femur (hip); 2. tibial shaft (shin bone); 3. ankle; 4. proximal humerus (shoulder); and 5: distal radius ( wrist)
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Go Fit Fast: Radiographic measurements, Patient related outcomes (PROs: PROMIS, HOOS, KOOS,), Loading/Activity pattern analysis | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  * Radiographic measurements
    o Healing (Radiographic Union Score in Tibia Fractures [RUST]/ Radiographic Union Score in Hip Fractures [RUSH])
  * Patient related outcomes
    * Patient Reported Outcome Measurement Information System (PROMIS): Physical Function (PF)/Pain Interference
    * Hip Disability and Osteoarthritis Outcome Score (HOOS) (assessing short- and long-term symptoms and function in hip injuries; the lower score indicates higher symptoms)
    * Knee Injury and Osteoarthritis Outcome Score (KOOS) (assessing short- and long-term symptoms and function in knee injuries; the lower score indicates higher symptoms)
  * Loading/Activity pattern analysis:
    * Number of steps with weight-bearing >80% body-weight (weight in kg)
    * pressure distribution [N/cm2]
    * center of pressure [mm]
    * ground reaction forces [N]
    * temporal and spatial parameters (time spent during gait [min], stance time [s], swing time [s], double support time [s], cadence [r/min], cycle time [s])
Recovery Trajectories PROMIS/Linking PROMIS: PROs: PROMIS, HOOS, KOOS, QuickDASH, FAAM | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PROs that measure physical limitations:
  * PROMIS PF (10 questions about physical function/mobility from self-care to strenuous activities; a higher score indicates a better self-reported capability)
  * PROMIS Upper Extremity (UE) (7 questions assessing arm and hand specific limitations, e.g. difficulty writing, lifting heavy objects; a higher score indicates a better function)
  * Disabilities of the Arm, Shoulder, and Hand (QuickDASH) (11 questions assessing outcomes in upper extremity disorders; a higher score indicates a greater disability)
  * HOOS
  * KOOS
  * Foot and Ankle Ability Measure (FAAM) (21 items of activities of daily living and 8 items on a Sports subscale. A higher score represent a higher level of physical function)
  * PROMIS Global Health (10 questions assessing physical health, mental health, and social health; a higher score indicates a better general health)

SECONDARY OUTCOMES:
PROMIS Pain Interference | from the treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PROMIS Pain Interference (8 questions) assesses the impact of pain on common activities of daily life including social, cognitive, emotional, physical, and recreational aspects. The higher score represents a higher pain level
PROMIS Depression | from the treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PROMIS Depression assesses negative mood (sadness, guilt), views of self (worthlessness, self-criticism) and diminished positive affect and engagement (loss of interest) within the previous week. The higher score represents higher depression level
PROMIS Anxiety | from the treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PROMIS Anxiety assesses levels of anxiety through measuring aspects of fear (e.g. fearfulness, feelings of panic), anxious misery (e.g. worry, dread), hyperarousal (e.g. tension, nervousness, restless) and some somatic symptoms related to arousal (e.g. dizziness). The higher score represent the higher level of anxiety
PROMIS Ability to Participate in Social Roles and Activities | from the treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PROMIS Ability to Participate in Social Roles and Activities item bank assesses the perceived ability to perform one's usual social roles and activities. The higher score represents better ability for social roles
Pain Self-Efficacy Questionnaire (PSEQ)-2 | from the treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PSEQ-2 assesses adaptive coping strategy and the confidence one can achieve one's goals in spite of pain. Items are scored on a 7-point Likert scale and added to form a total score ranging from 0 to 12, with higher scores indicating greater self-efficacy
Patient Activation Measure (PAM)-10 | from the treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PAM-10 assesses activation and the personal and psychological competencies. PAM segments individuals into one of four activation levels along an empirically derived 100-point scale. Individuals in the highest activation level are proactive with their health, have developed strong self-management skills, and are resilient in times of stress or change.
Cognitive assessment | Pre-treatment
  The MiniCog is a 3-minute instrument assessing cognitive impairment. It consists of two components, a 3-item recall test for memory and a simply scored clock drawing test. A total score ranges from 0 to 5. A score of zero, one or two out of five points in total, indicates a concern in cognitive functioning.
Mobility Scores | Pre-treatment
  Parker Mobility Scale assess the patient's ability to perform indoor walking, outdoor walking, and shopping before the fracture. A score ranges between 0 and 3 (0 = not at all, 1 = with help from another person, 2 = with an aid, and 3 = no difficulty and no aid) for each function, resulting in a total score ranging from 0 (no walking ability at all) to 9 (fully independent).

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Heng, Principal Investigator — Massachusetts General Hospital Harvard Orthopaedic Trauma Initiative; Prakash Jayakumar, Principal Investigator — Dell Medical School, University of Texas at Austin; Tim Pohlemann, Principal Investigator — Saarland University Hospital
Locations (15):
- United States (4):
  - Cedars-Sinai Department of Orthopaedics, Los Angeles, California
  - University of Miami, Jackson Memorial Hospital Ryder Trauma Center, Miami, Florida
  - Massachusetts General Hospital Harvard Orthopaedic Trauma Initiative, Boston, Massachusetts
  - The Value Institute / Department of Surgery and Peri-operative Care. Dell Medical School, University of Texas at Austin, Austin, Texas
- Univ.-Klinik für Orthopädie und Traumatologie, Innsbruck, Austria
- Fundación Santa Fe de Bogotá, Bogotá, Colombia
- Germany (5):
  - Centrum für Muskuloskeletale Chirurgie (CMSC) Charite - Universitätsmedizin Berlin, Berlin
  - University Hospital Freiburg, Freiburg im Breisgau
  - Saarland University Hospital Department of Trauma, Hand and Reconstructive Surgery, Homburg
  - Institut für Biomechanik Berufsgenossenschaftliche Unfallklinik Murnau, Murnau am Staffelsee
  - Abteilung für Unfall- und Wiederherstellungschirurgie BG Klinik Tübingen, Tübingen
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Isala Clinics, Zwolle
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No